CLINICAL TRIAL: NCT03813329
Title: The Effects of a Novel Bicarbonate Loading Protocol on Elite Running Performance. A Randomized Placebo-controlled Trial
Brief Title: Effects of Novel Sodium Bicarbonate Ingestion of Buffering Capacity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Long Island University (Other)
Collaborators: California State University, Los Angeles (Other)
Responsible Party: Principal Investigator, Amerigo Rossi, Assistant Professor, Long Island University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Rossi01
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: PERFORMANCE-ENHANCING EFFECT
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Opaque gelatin capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 4 progressively larger doses (110 mg·kg-1 - 200 mg·kg-1) of Calcium carbonate
  Interventions: Dietary Supplement: Modified Sodium Bicarbonate; Dietary Supplement: Acute Sodium Bicarbonate; Dietary Supplement: Calcium carbonate (placebo)
- Acute Sodium Bicarbonate (Active Comparator): 3 doses of calcium carbonate (110 mg·kg-1, 130 mg·kg-1, 160 mg·kg-1), followed by one acute does (300 mg·kg-1) of sodium bicarbonate.
  Interventions: Dietary Supplement: Modified Sodium Bicarbonate; Dietary Supplement: Acute Sodium Bicarbonate; Dietary Supplement: Calcium carbonate (placebo)
- Modified Sodium Bicarbonate (Experimental): 4 progressively larger doses (110 mg·kg-1 - 200 mg·kg-1) of sodium bicarbonate
  Interventions: Dietary Supplement: Modified Sodium Bicarbonate; Dietary Supplement: Acute Sodium Bicarbonate; Dietary Supplement: Calcium carbonate (placebo)

INTERVENTIONS:
Dietary Supplement: Modified Sodium Bicarbonate — 4 progressively larger doses (110 mg·kg-1 - 200 mg·kg-1) of sodium bicarbonate
Dietary Supplement: Acute Sodium Bicarbonate — 3 progressively larger doses of calcium carbonate followed by one acute dose of sodium bicarbonate (300 mg/kg)
Dietary Supplement: Calcium carbonate (placebo) — 4 progressively larger doses (110 mg·kg-1 - 200 mg·kg-1) of calcium carbonate

SUMMARY:
One purpose of the present study was to evaluate the effect of elevating serum bicarbonate concentration more than had been achieved in previous studies without inducing potentially ergolytic GI distress. In order to do so, a modified SB ingestion protocol (ModSB) of 4 progressively larger doses (110 mg·kg-1 - 200 mg·kg-1) was administered. It was hypothesized that ModSB would significantly elevate serum bicarbonate concentration to a greater extent than would an acute SB ingestion protocol (AcuteSB).

This study was also designed to corroborate the results of previous studies regarding the ergogenic effects of sodium bicarbonate ingestion. Most studies have administered sodium bicarbonate in solutions, which would make the participants aware of the substance ingested due to the distinctive flavor of SB, possibly inducing a placebo effect. All doses in the present study were administered in gelatin capsules to mask the flavor of the ingested substances, maintaining participant blindness to the procedure.

Blood samples were collected at baseline and following placebo (CaCO3), acute sodium bicarbonate ingestion, and modified sodium bicarbonate ingestion to determine the effects of the ingestion protocols on serum bicarbonate, sodium and lactate concentrations, as well as on serum pH and blood hematocrit. The study design was a randomized double-blind crossover.

ELIGIBILITY:
Inclusion Criteria:

* Peak oxygen consumption greater than 60 ml·kg-1·min-1 (men) or 50 ml·kg-1·min-1 (women)
* Currently training; defined as at least 5 days·week-1 of running
* Elite-level performance (750 or more points on the International Associations of Athletics Federations Scoring Table) for an 800m-5000m race during the preceding 6 months.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-05-01 (Actual); Primary Completion 2004-10-31 (Actual); Study Completion 2005-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration of serum sodium bicarbonate (mmol·L-1) | 24 hours
  Blood was drawn via venipuncture and allowed to coagulate at room temperature for 25 minutes and then spun in a refrigerated centrifuge for 10 minutes. The serum was pipetted into three small vials.
  One vial was tested for bicarbonate concentration in duplicate with a carbon dioxide liquid stable reagent method (TR28321, Thermo Electron Corporation, Waltham, MA) using a spectrophotometer (Lambda 20, PerkinElmer, Waltham, MA).

SECONDARY OUTCOMES:
Concentration of serum sodium (mmol·L-1) | 24 hours
  Blood was drawn via venipuncture and allowed to coagulate at room temperature for 25 minutes and then spun in a refrigerated centrifuge for 10 minutes. The serum was pipetted into three small vials.
  One vial was analyzed for sodium concentration (Vitros DT60 II, Ortho-Clinical Diagnostics, Rochester, NY)
pH | 24 hours
  The serum in one vial was immediately analyzed for pH using the Orion 720A+ (Thermo Electron Corporation, Waltham, MA)
Blood hematocrit (%) | 24 hours
  Blood was drawn via venipuncture. Two capillary tubes were immediately filled from the blood samples to be tested for hematocrit via the microhematocrit method.
Likert scale for self-reported gastrointestinal distress (1-10) | 24 hours
  Gastrointestinal distress was assessed via self-report on a Likert scale of 1-10.

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Marcus A, Rossi A, Cornwell A, Hawkins SA, Khodiguian N. The effects of a novel bicarbonate loading protocol on serum bicarbonate concentration: a randomized controlled trial. J Int Soc Sports Nutr. 2019 Sep 18;16(1):41. doi: 10.1186/s12970-019-0309-4. PMID 31533750